CLINICAL TRIAL: NCT04623749
Title: Percutaneous Versus Endoscopic Guided Fine Needle Aspiration Cytology in Diagnosis of Pancreatic Masses
Brief Title: Percutaneous Versus EUS FNAC in Pancreatic Masses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ola Kamal Mohammed Galal (Other)
Responsible Party: Sponsor-Investigator, Ola Kamal Mohammed Galal, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNAC in pancreatic masses
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Neoplasm; Pancreatic Cyst; Pancreatic Abscess
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous US guided FNAC in pancreatic masses (Active Comparator)
  Interventions: Procedure: US
- EUS guided FNAC in pancreatic masses (Active Comparator)
  Interventions: Procedure: EUS

INTERVENTIONS:
Procedure: US — Percutaneous Ultrasound guided FNAC
  Arms: Percutaneous US guided FNAC in pancreatic masses
Procedure: EUS — Endoscopic Ultrasound guided FNAC
  Arms: EUS guided FNAC in pancreatic masses

SUMMARY:
We aim to evaluate the role of Ultrasound-guided (USG) fine needle aspiration cytology (FNAC) in diagnosis of pancreatic masses compared to endoscopic ultrasound (EUS) guided fine needle aspiration cytology (FNAC).

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related mortality in the United States. Over 45,000 patients are diagnosed each year in the United States, and the majority of these patients succumb to their disease. Eighty percentages of patients are diagnosed with advanced, unrespectable disease. According to the latest statistics, only 7 % of patients survive 5 years after diagnosis. While the 5-year survival rate improves to 25 % in patients presenting with stage 1or localized disease, only 9 % of patients are identified at this early stage. The majority of patients (53%) presents with distant metastatic disease, and have a 5-year survival of 2%.

Improving the prognosis of patients with pancreatic cancer is a challenge. Overall, pancreatic cancer has one of the worst prognoses among all cancers; however, the prognosis is better if cancer is detected at an early stage. For example, patients with pancreatic cancers ≤1 cm in size at the time of diagnosis have a 5-year survival rate of 80.4% . Because such small cancers now account for 0.8% of all pancreatic cancer, detection of more small cancers would contribute to improving mortality rates.

The diagnostic approach to a possible pancreatic mass lesion relies first upon various non-invasive imaging modalities, including computed tomography, ultrasound, and magnetic resonance imaging techniques. Once a suspect lesion has been identified, tissue acquisition for characterization of the lesion is often paramount in developing an individualized therapeutic approach. Tools , in addition to radiologic imaging , currently employed in the initial evaluation of a patient with a pancreatic mass lesion include serum tumor markers , endoscopic retrograde cholangiopancreatography, Ultrasound-guided (USG) fine needle aspiration cytology (FNAC) and endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) .

Advancements in radiologic and endoscopic ultrasound (EUS) imaging have improved our ability to detect and stage pancreatic masses allowing for more selective surgical intervention for patients with resectable disease. Owing to the low sensitivity of cross-sectional imaging to detect small tumors in the pancreas.

Endoscopic ultrasound (EUS), in which the tip of the endoscope contains a high-frequency transducer , provides high resolution images of the pancreas. Indeed , its high resolution in experienced hands enables detection of focal lesions as small as 2-5 mm .

Ultrasound-guided (USG) fine needle aspiration cytology (FNAC) has emerged as a primary diagnostic modality in investigation in patients with pancreatic lesions. This technique was introduced into clinical practice nearly 3 decades ago and has proved to be a simple, cost-effective and minimally invasive technique that can yield material for tissue diagnosis .

ELIGIBILITY:
Inclusion Criteria:

* 50 Patients in different sex & age groups with pancreatic masses

Exclusion Criteria:

* Any general contraindications for FNAC or EUS in some cases as Coagulopathy with INR >1.5 or platelet count <50,000/mmc, Antithrombotic therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Yield, as defined by the percentage of patients in whom a histologically interpretable specimen will be retrieved by Trans abdominal US-FNAC. diagnostic accuracy | intraopeatve
  Percutaneous US guided FNAC technique

SECONDARY OUTCOMES:
Yield, as defined by the percentage of patients in whom a histologically interpretable specimen will be retrieved by EUS-FNAC. diagnostic accuracy | intraoperative
  EUS guided FNAC technique

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Egawa S, Toma H, Ohigashi H, Okusaka T, Nakao A, Hatori T, Maguchi H, Yanagisawa A, Tanaka M. Japan Pancreatic Cancer Registry; 30th year anniversary: Japan Pancreas Society. Pancreas. 2012 Oct;41(7):985-92. doi: 10.1097/MPA.0b013e318258055c. PMID 22750974
- See also: Related Info — http://ganjoho.jp/en/professional/statistics/brochure/2017_en.html
- See also: Related Info — http://seer.cancer.gov/csr/1975_2015/